CLINICAL TRIAL: NCT05391503
Title: A Circadian Medicine Light-based Intervention for Obsessive-compulsive Disorder (OCD)
Brief Title: Light Therapy for Obsessive-compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Rebecca Cox, Postdoctoral fellow, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 270-FP-22
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: circadian; sleep; anxiety; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Active Comparator): Active light therapy
  Interventions: Behavioral: Light therapy
- Control treatment (Placebo Comparator): Placebo light therapy
  Interventions: Behavioral: Placebo light therapy

INTERVENTIONS:
Behavioral: Light therapy — Morning bright light for 60 minutes after awakening
  Arms: Active treatment
Behavioral: Placebo light therapy — Placebo morning bright light for 60 minutes after awakening
  Arms: Control treatment

SUMMARY:
The purpose of this study is to examine the effect of a light-based circadian treatment on OCD symptoms in adults with OCD and late bedtimes. This study will have important implications for understanding the role of circadian rhythms in the etiology and treatment of OCD.

DETAILED DESCRIPTION:
Prior to the start of this study, there are screening procedures to ensure participants meet the criteria for the study. At the first consent screening appointment, participants will learn more about the study and answer questionnaires. All of the results of the screening procedures are confidential and will only be used by the study staff to determine eligibility for the study.

This study is 5 weeks long and involves 4 in-person lab visits at the Sleep and Chronobiology Lab. Participants will be randomly assigned to either an active or placebo light therapy treatment condition. Visit 1 will involve additional screening to determine eligibility, including questionnaires and interviews. If eligible, participants will then track their sleep for 2 weeks at home with a wrist-worn activity monitor and a sleep diary. Visit 2 will take place in the lab from 5:30pm until 1 hour after participants typical bedtime. The investigators will ask participants to provide saliva samples hourly to measure melatonin and complete questionnaires. The investigators will provide treatment instructions at this visit. Investigators will then ask participants to engage in the treatment at home for 3 weeks. Investigators will schedule 1 in-person visit (Visit 3) and 1 phone call to assess adherence to the treatment during these 3 weeks. Visit 4 will take place in the lab after the treatment is finished. Visit 4 will last from 5:30pm until 1.5 hours after participants typical bedtime and will involve hourly saliva samples to measure melatonin, questionnaires, and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Primary OCD diagnosis (according to the Diagnostic and Statistical Manual of Mental Disorders 5)
* Bedtime 0100 or later
* Age 18-35
* English speaking

Exclusion Criteria:

* Subjects must not be currently participating in another research study that would influence their participation in our study.
* Past 6-month substance use disorder
* Lifetime psychosis or bipolar disorder
* Current sleep disorder (DSWPD and insomnia excepted)
* Significant, active suicidal ideation or behaviors in the past 6 months
* Intellectual disability
* Engaged in evidence-based psychotherapy for OCD
* History of light therapy or cognitive behavior therapy for insomnia
* Night shift work or travel outside of Mountain Standard Time in the past month
* Pregnant, trying to become pregnant, or breastfeeding
* Change in psychotropic medication in the past month
* Prescribed or over the counter sleep medication use in the past month
* Beta-block or monoamine oxidase inhibitor use in the past month

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Obsessive-Compulsive Inventory-Revised score | 3 weeks
  Self-reported OCD symptoms. Minimum score=0, maximum score=74. Higher scores indicate worse outcome

SECONDARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale score | 5 weeks
  Interviewer-assessed OCD symptoms. Minimum score=0, maximum score=40. Higher scores indicate worse outcome

OTHER OUTCOMES:
Circadian phase | 3 weeks
  Circadian phase assessed by dim light melatonin onset (DLMO)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Cox, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Sleep and Chronobiology Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data generated from the proposed work that is presented in a peer reviewed journal will be de-identified.
  Other data that is presented in a peer reviewed journal will be archived indefinitely and made available upon request.